CLINICAL TRIAL: NCT02625194
Title: The Utility of Oxygen Insufflation During Flexible Fiberoptic Bronchoscope-guided Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2015-0218
Record Dates: First submitted 2015-11-25; First posted 2015-12-09 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Experimental): Oxygen is supplied through suction port in bronchoscope during bronchoscope-guided intubation.
  Interventions: Drug: Oxygen
- Control (No Intervention): Bronchoscope-guided intubation is performed without oxygen supply.

INTERVENTIONS:
Drug: Oxygen — Oxygen is supplied through suction port during bronchoscope-guided intubation.
  Arms: Oxygen

SUMMARY:
This study investigate the utility of continuous oxygen insufflation during fiberoptic bronchoscope-guided intubation.

One group receives oxygen via suction channel of fiberoptic bronchoscope during intubation.

The other group does not receive oxygen during fiberoptic bronchoscope-guided intubation.

Then, the velocity of deoxygenation difference of PaO2(baseline

DETAILED DESCRIPTION:
Fiberoptic bronchoscope-guided intubation is a gold standard for intubation of a patient with anticipating difficult airway. This technique takes several minutes without oxygen supply, which results in hypoxia when it prolonged. If continuous supply of oxygen during procedure improve the oxygenation, we can reduce the risk of hypoxemia and increase the safety margin during procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients who have surgery under general oral endotracheal anesthesia with invasive arterial blood pressure monitoring

Exclusion Criteria:

* history of lung disease
* abnormality in chest x-ray
* anticipating difficult intubation
* pregnant women
* who is unable to understand and agree the consent form

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Velocity of PaO2 decrease | from mask removal to 1st manual ventilation after intubation, up to 5 minute
  After administration of anesthetic agents and manual ventilation of 5 minutes, arterial blood sampling is collected. Then bronchoscope-guided intubation performed and arterial blood sample is collected immediately after the intubation completed. Time for intubation (between 1st and 2nd blood sample) is recorded. The difference of PaO2(before & after intubation) is divided by the time taking for intubation.

SECONDARY OUTCOMES:
success of intubation | 300 sec after the beginning of intubation
  After 1st trial of intubation, the success of intubation is recorded. If it takes more than 300 sec, it will be considered failure.
PaO2 | 1. 5 minutes after manual ventilation / 2.right before 1st manual ventilation after intubation, up to 5 minute
  arterial blood samples are collected before and after intubation.
PaCO2 | 1. 5 minutes after manual ventilation / 2.right before 1st manual ventilation after intubation, up to 5 minute
  arterial blood samples are collected before and after intubation.
pH | 1. 5 minutes after manual ventilation / 2.right before 1st manual ventilation after intubation, up to 5 minute
  arterial blood samples are collected before and after intubation.
visual field | throughout the intubation with bronchoscope, upto 5 minute
  Visual field is evaluated by the blinded observer. It is evaluated as followed;excellent, good, poor, impossible

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Soo Lee, MD, Study Chair — Yonsei University Gangnam Severance Hospital
Locations (1):
- Gangnam severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Roh GU, Kang JG, Han JY, Chang CH. Utility of oxygen insufflation through working channel during fiberoptic intubation in apneic patients: a prospective randomized controlled study. BMC Anesthesiol. 2020 Nov 10;20(1):282. doi: 10.1186/s12871-020-01201-9. PMID 33167909